CLINICAL TRIAL: NCT01362842
Title: Psychological and Physical Distress and Care Needs in Operable Lung Cancer Patients Receiving Surgery
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Other Study IDs: NTUH-201012108RC
Record Dates: First submitted 2011-05-27; First posted 2011-05-30 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2010-12

CONDITIONS: Anxiety Postoperative; Patient Non-Compliance; Psychological Distress
Keywords: Lung Cancer; Symptom distress; Post-operation; Anxiety; Depression; Uncertainty; Fear of recurrence; Self-efficacy; Needs
MeSH Terms: conditions — Patient Compliance; Lung Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The lung cancer is the most has the life minacity in all kinds of cancers, and it also remains the most common cause of cancer-related death in the world. The group of lung cancer patients are suffer from huge disease impact that came from high mortality. Not only the course of treatment that patients has been diagnosis through operation is more faster, but also those who could be capable of operated are stabilized to keep follow-up at out-patient clinic. But in the next following five years after operation, they may take different dysfunctional level or some kinds of symptom distress. The effect has a great influence on those patients that have to face extended emotional impact, symptom distress and life style change. In addition, most of them concern about recurrent all the time in the remission. These situation needs us to place importance on it.

The purposes of this study are to investigate psychological and physical distress and care needs in operable lung cancer patients receiving surgery. This survey includes two parts of physical and mental condition. First, the investigators are scoring their symptom severity and quality of life to check physical condition. Seconded, the mental condition will use validated questionnaires to realize the relationship of anxiety, depression, uncertainty, fear of recurrence, self-efficacy and needs. Final, compare all of the data to patients' needs.

This study is a cross-sectional designs with convenience sampling that conform to the investigators recruited requirements. The investigators will recruit from the clinic of thoracic surgery in one medical center in Taipei and take five structured requirements. And the investigators are going to collect data from January, 2011 to December, 2012. Also expect results are lung cancer outpatients after surgery that more physical dysfunction or more depress of mental condition, it will lead patients' needs increased or significant difference. In conclusion, this study analyzes their needs in the remission that consequences can be medical professionals' reference material.

DETAILED DESCRIPTION:
Inclusion Criteria:

lung cancer patients after surgery stage I, II and IIIA surgery for 3 months to 5 years over 20 years old

Exclusion Criteria:

lung cancer recurrence conscious unclear and do not know having cancer used to be treat (surgery, chemotherapy or radiotherapy) in 3 months. be uncomfortable or cooperate to fill the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer patients after surgery
* stage I, II and IIIA
* surgery for 3 months to 5 years
* over 20 years old

Exclusion Criteria:

* lung cancer recurrence
* conscious unclear and do not know having cancer
* used to be treat (surgery, chemotherapy or radiotherapy) in 3 months.
* be uncomfortable or cooperate to fill the questionnaire.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thoracic surgery outpatients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yeur-Hur Lai, Ph. D., Study Chair — Department of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hosptial, Taipei, Taiwan